CLINICAL TRIAL: NCT04287257
Title: Pulsed Electromagnetic Fields in the Treatment of Fresh Distal Radius Fractures. A Prospective, Double Blind, Placebo Controlled, Randomized Trial
Brief Title: PEMF in the Treatment of Fresh Distal Radius Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of Research and Developement Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0597-19-TLV
Record Dates: First submitted 2020-02-18; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment + Active FHP (Active Comparator): The PEMF device - FHP (supplied by commercial support) will be placed under the cast in the ER after diagnosing the fracture and will be applied for 24 hours a day continuously for 30-40 days.
  Interventions: Device: Fracture Healing Patch (FHP)
- Standard treatment + Sham FHP (Sham Comparator): Half of the PEMF devices will be not activated at random before the application to the patients. Two types of activators will be provided by the company: active and sham. Sham activated devices will give outward signs of normal function but will not generate a signal. The investigators will be unaware of the device's functionality. The patients will not be able to determine whether the device is working or not. At study completion, device serial numbers will be used to determine which patients received a working device. The company supplying the PEMF-devices will have no knowledge of patient outcome.
  Interventions: Device: Fracture Healing Patch (FHP)

INTERVENTIONS:
Device: Fracture Healing Patch (FHP) — The Fracture Healing Patch (FHP) is an external silicone patch that contains inside micro-electronic modulus, which generates a pulsed electromagnetic field (PEMF) to enhance and improve fracture healing. The FHP is placed under the cast at the fracture site. Throughout the treatment period the FHP produces a pulsed electromagnetic field. The FHP houses a battery, a microelectronic module and a coil that produce the PEMF.

SUMMARY:
Distal radial fractures (DRF) are the most common fractures encountered in health care. Annualized estimates in the United States alone suggest an incidence of approximately 640,000 cases, and rising, per year. Most fractures may be treated in a plaster cast, but unstable fractures tend to displace without a surgical procedure. 1

Pulsed electromagnetic field (PEMF) is one modality commonly used to stimulate bone generation throughout various clinical settings including orthoapedic surgery. PEMF has been shown to primarily effect vascular generation, formation and neovascularization2,3. This may help decrease time to healing and allow patients to return to normal activities sooner.

Additional study demonstrated that PEMF exposure increased cell proliferation, adhesion and the osteogenic commitment of MSCs, even in inflammatory conditions. In this in-vitro model PEMFs increased the expression of anti-inflammatory cytokines, such as IL-10, and reduced the expression of the pro-inflammatory cytokine IL-1 4.

The distal radius fracture was chosen as the model to test the effects of PEMF treatment because it includes both trabecular and cortical bone, is accessible for radiographs, has little soft tissue that can distort the radiograph, and is amenable to multiple functional endpoints.

The purpose of the study is to determine whether the use of FHP by means of pulsed electromagnetic fields in acute distal radius fractures will accelerate healing both clinically and radiotralogically

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with closed unilateral dorsally angulated fracture of the distal radius (Colles') visible by x-ray.
2. Subjects treated conservatively by immobilization ± closed reduction
3. Age >18 years
4. Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.

Exclusion Criteria:

1. Subjects with intra articular fracture or extra-articular fracture that meets the criteria for operative fracture fixation.
2. Subjects with pins or plates in the wrist
3. Sustained previous fractures or bone surgery in the currently fractured distal forearm
4. Synovial pseudarthrosis
5. Subjects with multiple trauma (several fractures at once)
6. Subjects suffering from joint diseases that affect the function of the wrist and/or hand of the injured arm.
7. Pregnancy
8. Women who are breast-feeding.
9. Women of childbearing potential and not using a medically accepted form of contraception when sexually active.
10. presence of a life supporting implanted electronical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in radiographic fracture healing | Radiographic images (X-ray) will be performed for each subject from day 0 and onward: week 2,4, 6 and 12.
  Change from baseline in radiographic fracture healing will be measured. Radiographic healing will be defined as the interval in days between the occurrence of the fracture and the time when bridging in three of four cortices is seen on X-ray images. A measurement will be made at each follow up evaluation by using Radius Union Scoring System (RUSS) score

SECONDARY OUTCOMES:
Change from baseline in improvement of function | Functional assessment will be performed at 4, 6 and 12 weeks from treatment
  For assessment of functional deficit, disability and pain level, the Patient Rated Wrist Evaluation (PRWE) will be used. The PRWE is an easy 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability.
  Pain Score = Sum of the 5 pain items (out of 50) Best Score = 0, Worst Score = 50 Function Score = Sum of the 10 function items, Divided by 2 (out of 50) Best Score = 0, Worst Score = 50 Computing the Total Score Total Score = Sum of pain + function scores Best Score = 0, Worst Score = 100

IPD SHARING:
Plan to Share IPD: No